CLINICAL TRIAL: NCT02683733
Title: The Efficacy and Tolerability of Bio-enhanced Curcumin (Diferuloylmethane) in the Induction of Remission in Patients With Mild to Moderate Ulcerative Colitis
Brief Title: Bio-enhanced Curcumin as an Add-On Treatment in Mild to Moderate Ulcerative Colitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rupa Banerjee, Consultant Gastroenterologist; Director, IBD Clinic, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIGINDIACurcumin1
Record Dates: First submitted 2016-02-10; First posted 2016-02-17 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Active Comparator): Patients will receive 5-Aminosalicylic acid as per their current treatment regimen and will also take Bio-enhanced curcumin twice daily after meals as per the following regimen:
  Starting dose: 50 mg BID of Bio-enhanced Curcumin Soft Gelatin Capsule Increase dose to 100 mg BID after two (2) weeks if there is no response to the drug
  Interventions: Dietary Supplement: Bio-enhanced Curcumin Soft Gelatin Capsule; Drug: 5-Aminosalicylic acid
- Control Arm (Placebo Comparator): Patients will receive 5-Aminosalicylic acid as per their current treatment regimen and will also take a placebo pill twice daily after meals
  Interventions: Drug: 5-Aminosalicylic acid

INTERVENTIONS:
Dietary Supplement: Bio-enhanced Curcumin Soft Gelatin Capsule — Each capsule is a bio-enhanced modification of curcumin (diferuloylmethane), which is a derivative of curcuma longa (rhizome extract)
  Other Names: Valdone
  Arms: Treatment Arm
Drug: 5-Aminosalicylic acid — Dosage is as instructed by patient's physician
  Other Names: 5-ASA

SUMMARY:
Inflammatory Bowel Disease, including ulcerative colitis, is thought to result from an imbalance of pro-inflammatory and anti-inflammatory factors. As such, the majority of treatment options are directed at attempting to control the chronic inflammation and prolonging remission of clinical symptoms. Several studies have proven that curcumin has well-established anti-inflammatory properties. However, curcumin has poor bioavailability and prior studies have needed to use high concentrations in order to study the efficacy of the product. The investigators propose that a bio-enhanced preparation of curcumin will require a lower dosage to reach and affect its target tissue and will subsequently produce less adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have mild to moderate ulcerative colitis, with a current Partial Mayo Index greater than or equal to 2 and less than or equal to 6
* Age 18 years and above
* Male or female
* Patients who have given consent and area able to follow the treatment given
* Patients who are able to record their responses in survey form at regular follow-up visits

Exclusion Criteria:

* Patients who are in remission from ulcerative colitis, or who have a Partial Mayo Index Score of 0 or 1
* Patients who have been taking azathioprine or mercaptopurine for <12 weeks for the treatment of their ulcerative colitis
* Patients who are taking steroids or biologic agents for the treatment of their ulcerative colitis
* Patients who have severe ulcerative colitis, or who have a Partial Mayo Index Score of 7 or above
* Patients who are noncompliant with medication or regular follow up visits
* Patients who are unable to or unwilling to record their responses in survey form
* Patients with comorbid illnesses, including: Diabetes Mellitus, Stage III or above Congestive Heart Failure, chronic pancreatitis, severe liver or renal disease
* Patients who have current gallstones or any biliary dysfunction
* Patients with anemia (Hemoglobin <10), thrombocytopenia, abnormal lymphocyte counts, or coagulation abnormalities
* Patients who currently have an ongoing severe infection/sepsis
* Patients with a history of malignancy
* Patients who are currently pregnant or nursing
* Patients who are current smokers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Time to induction of clinical remission in the treatment arm compared with time to induction of clinical remission in control arm | 1 year
  Clinical remission is recorded by a Partial Mayo Index score of 0-1
Time to induction of endoscopic remission in the treatment arm compared with time to induction of endoscopic remission in control arm | 1 year
  Endoscopic remission is defined as endoscopic mucosal healing, is recorded by Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score of <3

SECONDARY OUTCOMES:
Percentage of patients in the treatment arm who experienced adverse events as compared with patients in the control arm | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rupa Banerjee, MD, DM, Principal Investigator — Asian Institutes of Gastroenterology
Locations (1):
- Asian Institutes of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee R, Pal P, Penmetsa A, Kathi P, Girish G, Goren I, Reddy DN. Novel Bioenhanced Curcumin With Mesalamine for Induction of Clinical and Endoscopic Remission in Mild-to-Moderate Ulcerative Colitis: A Randomized Double-Blind Placebo-controlled Pilot Study. J Clin Gastroenterol. 2021 Sep 1;55(8):702-708. doi: 10.1097/MCG.0000000000001416. PMID 32889959